CLINICAL TRIAL: NCT04956666
Title: A Multicentre, Roll-over Study to Provide Continued Treatment With Lyophilized Pegaspargase (S95014) in Pediatric Patients With Acute Lymphoblastic Leukemia (ALL)
Brief Title: A Roll-over Study to Provide Continued Treatment With Lyophilized Pegaspargase (S95014) in Pediatric Patients With Acute Lymphoblastic Leukemia (ALL)
Acronym: ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry); Les Laboratoires Servier (L.L.S), Russia (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL2-95014-003; 2020-004895-17 (EudraCT Number)
Record Dates: First submitted 2021-06-18; First posted 2021-07-09 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Phase II; Oncology / Haematology; Continued treatment; Pegaspargase; Lyophilized pegaspargase; Roll-over study / extension study
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lyophilized S95014 (Experimental): Lyophilized S95014 reconstituted was provided 5 mL of extractable volume with the concentration of 750 U/mL.
  The vial of lyophilized powder (3.750 U/vial) was reconstituted with 5.2 mL of Sterile Water For Injection to obtain a 750 U/mL solution for single use.
  Interventions: Drug: Lyophilized S95014

INTERVENTIONS:
Drug: Lyophilized S95014 — Each patient was administrated, over 1 to 2 hours, every 2 weeks Lyophilized S95014 intravenously at the dose of 1000, 2000 or 2500U/m2, as per investigator's judgement.
  In total, 9 infusions of lyophilized S95014 were administrated (at week 7, 9, 11, 15, 17, 19, 23, 25 and 27).Patients received other backbone chemotherapy agents as per ALL-MB 2015.

SUMMARY:
The purpose of this study is to provide treatment with lyophilized S95014 in pediatric patients with ALL who completed the CL2-95014-002 study during the induction phase and who are clinically benefitting from S95014 without major toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient who completed the CL2-95014-002 study
* Patient currently receiving clinical benefit from previous treatment with S95014 as per investigator's judgment
* Signed informed consent and assent, when appropriate
* Highly effective contraception method

Non-inclusion Criteria:

* Unlikely to cooperate in the study
* Pregnant and lactating women
* Participant already enrolled in the study (informed consent signed)
* Prior surgery or bone marrow transplant related to the studied disease
* History of sensitivity to polyethylene glycol (PEG) or PEG-based drugs
* Psychiatric illness/social situation that would limit compliance with study requirements
* Group "E" and "T-HR" patients according to ALL-MB 2015 protocol classification
* Major safety issue due to previous S95014 administration (e.g. non recovery of safety parameters, serious hypersensitivity, serious pancreatitis, serious haemorrhage, serious thromboembolic event)
* Significant laboratory abnormality or uncontrolled intercurrent illness (e.g. life-threatening acute tumor lysis syndrome, symptomatic congestive heart failure, cardiac arrhythmia, severe or uncontrolled active acute infection) likely to jeopardize the patients' safety or to interfere with the conduct of the study, in the investigator's opinion

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Isaakovich Karachunskiy, PhD, Principal Investigator — Director of Institute of Oncology, Radiology and Nuclear Medicine. Dmitry Rogachev National Medical Research Center of Pediatric Hematology, Oncology and Immunology
Locations (6):
- Russia (6):
  - Regional Children Clinical Hospital, Chelyabinsk
  - Children Regional Clinical Hospital, Krasnodar
  - Russian Children Clinical Hospital, Moscow
  - Regional Children Hospital, Nizhny Novgorod
  - V.A. Almazov National Medical Research Center, Saint Petersburg
  - Regional Children Clinical Hospital, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH).The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com
- Available data/document: Study Protocol — https://clinicaltrials.servier.com
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Lyophilized S95014: Lyophilized S95014 reconstituted provided 5 mL of extractable volume with the concentration of 750 U/mL.
Period: Overall Study
Arm/Group | Lyophilized S95014
Started | 75 (One patient, included here in the 75 that started the study, dropped out before treatment due to the investigator's decision of a change in treatment strategy. Therefore, a total of 74 patients were treated and analyzed. This patient was also included in the "reason not completed" "physician decision" count.)
Completed | 52
Not Completed | 23
Not completed — Adverse Event | 18
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Groups:
- Lyophilized S95014: Lyophilized S95014 reconstituted was provided 5 mL of extractable volume with the concentration of 750 U/mL.
Arm/Group | Lyophilized S95014
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (3.83)
Age, Customized [Count of Participants; unit: Participants]
  Age Category: < 10 years | 60
  Age Category: [10, 15] years | 12
  Age Category: ≥ 16 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 71
  Race: Asian | 2
  Race: Multiple | 1
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status scores range from 0 to 5, with 0 being fully active and 5 being dead, and are graded by the investigator during the participants clinical examination.
  Participants
    ECOG Performance Status: 0 | 14
    ECOG Performance Status: 1 | 46
    ECOG Performance Status: 2 | 14
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 16.45 (3.51)
Body Surface Area (m^2) [Mean (Standard Deviation); unit: m^2] | 0.902 (0.356)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs) (Safety and Tolerability)
Description: All Adverse events (AEs) including Treatment Emergent Adverse Events (TEAEs) causality and severity based on NCI CTCAE 5.0.
Time Frame: Through study completion, approximately 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lyophilized S95014
Number analyzed (Participants) | 74
Participants
  Number of Participants with an Adverse Event | 74
  Number of Participants with an Treatment Emergent Adverse Event | 74
  Number of Participants with a Grade 3 or 4 Treatment Emergent Adverse Event | 72
  Number of Participants with a Serious Treatment Emergent Adverse Event | 27

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 19 months
Description: Throughout the study multiple safety visits were conducted and patients underwent physical examinations, electrocardiograms, hematology, blood biochemistry, coagulation parameters, urinalysis, hepatitis serology, cardiac imaging, and vital sign measurements. During these assessments any abnormal values, test or exam results constituted an adverse event if they meet criteria or were deemed clinically significant by the investigator.
Arm/Group | Lyophilized S95014
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 27/74
Other Adverse Events (participants affected / at risk) | 68/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lyophilized S95014 (N=74)
Hypersensitivity (Immune system disorders) | 11
Anaphylactic reaction (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 3
COVID-19 pneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Neutropenic sepsis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis gangrenous (Infections and infestations) | 1
Device related bacteraemia (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Agranulocytosis (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Ejection fraction decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
General physical health deterioration (General disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lyophilized S95014 (N=74)
Antithrombin III decreased (Investigations) | 53
Neutropenia (Blood and lymphatic system disorders) | 46
Blood fibrinogen decreased (Investigations) | 48
Alanine aminotransferase increased (Investigations) | 35
Anaemia (Blood and lymphatic system disorders) | 32
Gamma-glutamyltransferase increased (Investigations) | 31
Aspartate aminotransferase increased (Investigations) | 24
Hypersensitivity (Immune system disorders) | 13
Leukopenia (Blood and lymphatic system disorders) | 20
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14
Protein S decreased (Investigations) | 12
Blood bilirubin increased (Investigations) | 11
Neutrophil count decreased (Investigations) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 11
COVID-19 (Infections and infestations) | 7
White blood cell count decreased (Investigations) | 8
Activated partial thromboplastin time prolonged (Investigations) | 7
Pyrexia (General disorders) | 7
Drug hypersensitivity (Immune system disorders) | 5
Lipase increased (Investigations) | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 5
Toxic neuropathy (Nervous system disorders) | 5
Blood albumin decreased (Investigations) | 4
Haemoglobin decreased (Investigations) | 4
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Ammonia increased (Investigations) | 3
Amylase increased (Investigations) | 3
Hyperammonaemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3
Lymphocyte count decreased (Investigations) | 3
Lymphopenia (Blood and lymphatic system disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Platelet count decreased (Investigations) | 3
Rhinitis (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT04956666/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT04956666/SAP_001.pdf